CLINICAL TRIAL: NCT07396129
Title: Assessing the Efficacy of High-Dose Lidocaine-Tetracaine Cream for the Treatment of Peripheral Neuropathic Pain: A Crossover Study in Elderly Patients Refractory to Pharmacological Treatments
Brief Title: Assessing the Efficacy of a High-Dose Lidocaine-Tetracaine Cream for the Treatment of Peripheral Neuropathic Pain
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 250502001
Record Dates: First submitted 2025-12-05; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-10

CONDITIONS: Neuropathic Chronic Pain
Keywords: neuropathic chronic pain; lidocaine; tetracaine; anesthetic cream; crossover study
MeSH Terms: interventions — Lidocaine; Tetracaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- All Participants, placebo cream (Placebo Comparator): In this crossover study, all the participants will take part as their own control group.
  Interventions: Drug: Placebo cream application
- All participants, active cream (Active Comparator): In this crossover study, all the participants will take part as their own control group.
  Interventions: Drug: Lidocaine (23%) + Tetracaine (7%)

INTERVENTIONS:
Drug: Lidocaine (23%) + Tetracaine (7%) — Application of the active cream (combination of both Lidocaine 23% / Tetracaine 7%) twice daily: once in the morning upon waking and once before sleep, for two weeks.
  Arms: All participants, active cream
Drug: Placebo cream application — (After a 30 day washout period) Application of the placebo cream twice daily under the same conditions as the active cream: once in the morning upon waking and once before sleep, for two weeks.
  Arms: All Participants, placebo cream

SUMMARY:
The goal of this clinical trial is to learn if the topical anesthetic cream works to treat neuropathic chronic pain in older adults who have not found sufficient relief undergoing other pain treatments and/or medications. The safety of this drug has already been tested in other studies. The main questions it aims to answer are:

* Does the anesthetic cream lower the pain of participants?
* Can the participants return to daily activities that they have quit due to chronic pain?
* What medical problems do participants have when using this cream?

Researchers will compare the anesthetic cream to a placebo (a look-alike substance that contains no drug) to see if it works to treat neuropathic chronic pain.

Participants will:

* Use the anesthetic cream or a placebo every day for 14 days
* Visit the clinic once every 2 weeks for checkups and tests
* Keep a diary of their symptoms and the number of times they use the anesthetic cream.

This study is divided into two phases, separated by 30 days.

* Phase 1: Application of the active cream (Lidocaine 23% / Tetracaine 7%) twice daily: once in the morning upon waking and once at night before bed.
* Phase 2: Application of the placebo cream under the exact same conditions.

The order of administration (active/placebo) will be randomly assigned.

Procedure: Participants will sign the informed consent form. A baseline evaluation will be conducted, assessing VAS (Visual Analog Scale) score, functionality, and quality of life.

The use of other medications will be recorded. The creams will be applied at home with weekly telephone follow-up and daily patient self-reporting. Evaluations will be conducted on day 14 of each phase. Follow-up controls will occur one and two months after the treatment is suspended. Adherence and adverse effects will also be logged.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older.
* Clinical diagnosis of peripheral neuropathic pain that has lasted for at least 6 months.
* Baseline Visual Analog Scale (VAS) pain score of 6 or higher.
* Ability to understand and sign the informed consent form.

Exclusion Criteria:

* Known hypersensitivity (allergy) to lidocaine, tetracaine, or any excipients (inactive ingredients) in the preparation
* Dermatological lesions (skin damage or sores) in the intended application area.
* Concomitant use of other topical therapies (creams, gels, patches) in the affected area.
* Severe cognitive impairment or unstable medical comorbidity.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-23 (Estimated)

PRIMARY OUTCOMES:
Reduction in pain (treatment area) | From Enrollment to the end of treatment at 2 months
  The Visual Analog Pain Scale, will be used to assess the reduction of pain, being 0 no pain and 10 the worst pain ever experienced.

SECONDARY OUTCOMES:
Better outcomes in daily function and quality of life | From enrollment to the end of treatment at 2 months
  The World Health Organization Disability Assessment Schedule scale: A tool used to measure overall disability and functioning across different life domains (e.g., cognition, mobility, participation).
  Every life domain will be asigned to a specific score in percentage:
  * 1% best case scenario, no disability and appropriate function.
  * 100% worst case scenario, fully dependent in most life domains.
Better outcomes in daily function and quality of life | From enrollment to the end of treatment at 2 months.
  EuroQol 5-Dimension 5-Level: A standardized instrument for measuring health-related quality of life.
  The participant will answer an every day task sheet, which will provide a specific score from 1 to 5:
  * being the best case scenario: no problem on completing the task.
  * 5 being the worst case scenario: not being able to complete the task.

IPD SHARING:
Plan to Share IPD: Undecided